CLINICAL TRIAL: NCT05612802
Title: A New Marker for Early Diagnosis of Pneumoperitoneum-Related Acute Kidney Injury: Insulin-Like Growth Factor-1 (IGF-1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Çağla Yazar, MD, Principal investigator, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KA22/178
Record Dates: First submitted 2022-09-06; First posted 2022-11-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury (Nontraumatic); Pneumoperitoneum
MeSH Terms: conditions — Acute Kidney Injury; Pneumoperitoneum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGF (Other): Creatinine and NGAL have been used successfully in the follow-up of acute kidney injury. In our study, in order to show the effect of pneumoperitoneum on acute kidney injury in patients scheduled for laparoscopic surgery, NGAL and IGF-1 values will be measured before, after and 24 hours after pneumoperitoneum, and these values will be compared.
  Interventions: Diagnostic Test: IGF-1

INTERVENTIONS:
Diagnostic Test: IGF-1 — We need to diagnose acute kidney injury in the early postoperative period. The markers examined so far do not provide enough information to diagnose acute kidney injury early. For this reason, many different biomarkers are used in the early diagnosis of acute kidney injury in many parts of the world. Thanks to our research, we can recognise the development of acute kidney injury at an early stage and determine whether a previously unused biomarker (IGF-1) is effective in the early diagnosis of acute kidney injury.

SUMMARY:
In our study, to show the effect of pneumoperitoneum on acute kidney injury in patients scheduled for laparoscopic surgery, NGAL and IGF-1 values will be measured before, after and 24 hours after pneumoperitoneum, and these values will be compared. In our study, we aimed to investigate the effect of pneumoperitoneum applied on acute kidney injury in patients who underwent laparoscopic surgery. Creatinine and NGAL have been used successfully in the follow-up of acute kidney injury. Our study investigates whether IGF-1 will be an effective indicator in acute kidney injury by comparing IGF-1 and NGAL values before pneumoperitoneum, after pneumoperitoneum and at the postoperative 24th hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years of both sexes
* ASA I-III Patients

Exclusion Criteria:

* Obesity,
* Chronic Kidney Disease,
* Chronic Renal Failure,
* Acute Renal Failure,
* Peripheral and ischemic vascular disease,
* Chronic Heart Failure,
* History of anaphylaxis,
* A-V block,
* Creatinine level >1.4,
* Neuromuscular disease,
* Malignant hypertension,
* Pyelonephritis,
* Urinary tract infectio,
* Severe inflammation/possible sepsis,
* Active malignancy,
* Patients with surgery reversion to laparotomy,
* Hemodynamic instability, need for vasopressors,
* Severe bleeding requiring blood transfusion,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute kidney injury in the early postoperative period with IGF-1 (insulin like growth factor-1) | before pneumoperitoneum, after pneumoperitoneum, and at the postoperative 24th hour.
  The researchers investigate whether IGF-1 will be an effective indicator in acute kidney injury by comparing IGF-1 and NGAL (Neutrophil gelatinase-associated lipocalin) values before pneumoperitoneum, after pneumoperitoneum and at the postoperative 24th hour.

CONTACTS AND LOCATIONS:
Overall Officials: NEDİM ÇEKMEN, PHD, Study Director — Baskent University
Locations (1):
- Çağla Yazar, MD, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gumbert SD, Kork F, Jackson ML, Vanga N, Ghebremichael SJ, Wang CY, Eltzschig HK. Perioperative Acute Kidney Injury. Anesthesiology. 2020 Jan;132(1):180-204. doi: 10.1097/ALN.0000000000002968. PMID 31687986
- [Background] Marton Filho MA, Alves RL, Nascimento PD Junior, Tarquinio GDS, Mega PF, Pinheiro Modolo NS. Effects of pneumoperitoneum on kidney injury biomarkers: A randomized clinical trial. PLoS One. 2021 Feb 19;16(2):e0247088. doi: 10.1371/journal.pone.0247088. eCollection 2021. PMID 33606739
- [Background] Sun B, Fu A, Wang R, Zhang Y. Influence of carbon dioxide pneumoperitoneum on the growth hormone-insulin-like growth factor I axis in mid- and late-pregnancy rats. J Obstet Gynaecol Res. 2015 Sep;41(9):1394-8. doi: 10.1111/jog.12734. Epub 2015 Jun 22. PMID 26098754
- [Background] Srisawat N, Kongwibulwut M, Laoveeravat P, Lumplertgul N, Chatkaew P, Saeyub P, Latthaprecha K, Peerapornratana S, Tiranathanagul K, Eiam-Ong S, Tungsanga K. The role of intraoperative parameters on predicting laparoscopic abdominal surgery associated acute kidney injury. BMC Nephrol. 2018 Oct 22;19(1):289. doi: 10.1186/s12882-018-1081-4. PMID 30348111